CLINICAL TRIAL: NCT06532539
Title: A Phase II, Single-arm, Multicenter Clinical Trial of Definitive Treatment With Cadonilimab, Paclitaxel, Cisplatin and Radiation for the Treatment of Locally Recurrent and Oligometastatic Endometrial Carcinoma
Brief Title: Cadonilimab With Chemoradiation for Recurrent and Oligometastatic Endometrial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Peng Xie, Director, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2024-160-01
Record Dates: First submitted 2024-07-22; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-06

CONDITIONS: Endometrial Neoplasms; Neoplasm Recurrence, Local; Neoplasm Metastasis
Keywords: Immunotherapy; Cadonilimab; Paclitaxel; Cisplatin; Radiation Therapy; Combined Modality Therapy; Clinical Trials, Phase II as Topic; Progression-Free Survival; Biomarkers, Tumor; Treatment Outcome; Safety
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Recurrence, Local; Neoplasm Metastasis; Neoplasms | interventions — TP protocol; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Chemotherapy：TP (Paclitaxel and Cisplatin) Immunotherapy：Cadonilimab Radiotherapy：All tumor lesions will be irradiated
  Interventions: Drug: Paclitaxel and Cisplatin; Drug: Cadonilimab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Paclitaxel and Cisplatin — Paclitaxel and Cisplatin Paclitaxel: 135 mg/m², intravenous infusion, Day 1, every 3 weeks (Q3W). Cisplatin: 75 mg/m², intravenous infusion, Days 1-3, every 3 weeks (Q3W). Duration: 6-8 cycles, until disease progression or intolerable adverse effects as judged by the investigator.
  Alternative: If contraindicated for cisplatin, or if there is an allergy to paclitaxel and/or cisplatin, alternative drugs such as different types of paclitaxel or carboplatin can be used.
  Other Names: TP
Drug: Cadonilimab — Cadonilimab: 5-10 mg/kg, intravenous infusion, Day 1, every 3 weeks (Q3W). Duration: Continuous administration until disease progression, death, intolerable toxicity, subject's voluntary withdrawal, investigator's decision for withdrawal, or a maximum of 24 months.
  Other Names: AK104
Radiation: Radiotherapy — Site Selection: Original site, lymph nodes, lung metastasis, bone metastasis, adrenal metastasis, brain metastasis, and other relatively isolated, well-vascularized lesions. Select at least one suitable lesion for radiotherapy based on the impact of the recurrent or metastatic lesion on the body, prioritizing lesions that cause symptoms, are life-threatening, or are expected to cause symptoms.All tumor lesions will be irradiated, which can be done in phases.
  Dosage and Fractionation: Conventional or hypofractionated radiotherapy, with a biologically effective dose (BED) of ≥ 72 Gy. Dose adjustments can be made for brain metastases.
  Timing: After completing relevant baseline examinations, radiotherapy can be implemented generally after 2-6 cycles of systemic therapy, or after the first cycle for small, solitary metastatic lesions.
  echnique: IMRT, TOMO, SBRT, 3D-BT, interstitial implantation therapy, or proton therapy.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of cadonilimab in combination with paclitaxel, cisplatin, and radiation therapy for the treatment of locally recurrent and oligometastatic endometrial carcinoma. The main questions it aims to answer are:

1. Does the combination therapy improve the overall response rate (ORR), progression-free survival (PFS), disease control rate (DCR), overall survival (OS), and safety in participants?
2. What are the predictive biomarkers of treatment efficacy, and how can this information better guide the use of immune-oncology drugs in combination therapy?

Participants will:

* Receive cadonilimab, paclitaxel, cisplatin, and radiation therapy according to a specified protocol.
* Visit the clinic for regular checkups and tests throughout the treatment period.
* Be monitored for and have records kept of ORR, PFS, DCR, OS, and safety.
* Provide hematologic and tissue samples to explore biomarkers.

This study will help determine if this combination therapy can become a new standard of care for patients with locally recurrent and oligometastatic endometrial carcinoma, as well as identify biomarkers to better guide treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. A written informed consent form must be signed before the implementation of any trial-related procedures.
2. Female, aged 18 years or older and 80 years or younger.
3. ECOG PS 0-1.
4. Newly diagnosed with histologically or cytologically confirmed primary endometrioid adenocarcinoma, serous carcinoma, clear cell adenocarcinoma, undifferentiated carcinoma, mixed cell adenocarcinoma, mesonephric adenocarcinoma, mucinous carcinoma, intestinal-type mesonephric-like adenocarcinoma, and carcinosarcoma, meeting the clinical diagnostic criteria for endometrial cancer.
5. Patients with locally recurrent or oligometastatic endometrial cancer after initial treatment. The number of recurrent and metastatic lesions is ≤5. Screening criteria for oligometastasis: lymph node metastases in the same region count as one metastatic lesion; liver metastases are limited to one; lung metastases are limited to three.
6. At least one site suitable for radiotherapy (including the primary lesion), measurable, and meeting the RECIST v1.1 criteria for evaluable lesions.
7. Tumor samples available for biomarker assessment.
8. Expected survival time ≥6 months.
9. Normal major organ function (within 7 days before enrollment), meeting the following criteria:

(1) Hematology standards (without blood transfusion or hematopoietic growth factor treatment within 14 days before enrollment):

1. Hemoglobin (HB) ≥80 g/L;
2. Absolute neutrophil count (ANC) ≥1.5×10^9/L;
3. Platelet count (PLT) ≥50×10^9/L; (2) No functional or organic diseases, meeting the following criteria:

a) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN, total serum bilirubin ≤1.5×ULN, alkaline phosphatase (ALP) ≤3×ULN, serum albumin ≥30 g/L; b) Serum creatinine (Cr) ≤1.5×ULN; if serum creatinine is >1.5×ULN, creatinine clearance (CrCl) ≥50 mL/min (calculated using the Cockcroft-Gault formula); c) Prothrombin time (PT) prolongation ≤6 seconds, activated partial thromboplastin time (APTT) ≤1.5×ULN; d) Thyroid-stimulating hormone (TSH) ≤ULN (if abnormal, FT3 and FT4 levels should be considered; if FT3 and FT4 levels are normal, enrollment is allowed); f) Left ventricular ejection fraction (LVEF) >50%. 11. Before starting the first treatment, all reversible toxic reactions from previous anti-tumor treatments must have resolved to ≤ grade 1 (based on CTCAE v5.0), excluding any grade of alopecia and pigmentation, ≤ grade 2 peripheral sensory neuropathy, and other abnormalities considered by the investigator and/or sponsor to pose a benefit-risk balance favoring the subject receiving the study treatment.

12. Non-surgically sterilized or childbearing potential female patients must use medically recognized contraception (e.g., intrauterine device, contraceptive pill, or condom) during the study treatment period and for 3 months after the end of the study treatment. Non-surgically sterilized childbearing potential female patients must have a negative serum or urine HCG test within 7 days before enrollment and must not be breastfeeding.

Exclusion Criteria:

1. Subjects with any active autoimmune disease or history of autoimmune disease (e.g., but not limited to: autoimmune hepatitis, interstitial lung disease, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or childhood asthma that has completely resolved and does not require any intervention in adulthood may be included; subjects with asthma requiring medical intervention with bronchodilators are not eligible).
2. Subjects currently using immunosuppressive agents or systemic, or absorbable local corticosteroid therapy to achieve immunosuppressive purposes (dose >10 mg/day prednisone or equivalent) and continuing use within 2 weeks prior to enrollment.
3. Known history of grade 3 or 4 immune-related adverse events associated with previous anti-tumor immunotherapy.
4. Poorly controlled cardiac clinical symptoms or diseases, such as: (1) NYHA class II or higher heart failure; (2) unstable angina; (3) myocardial infarction within the past six months; (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; (5) QTc >450 ms (males); QTc >470 ms (females).
5. Coagulation dysfunction (INR >1.5 or PT >16 s), bleeding tendency, or receiving thrombolytic or anticoagulant therapy.
6. Subjects who have received radiotherapy, chemotherapy, hormone therapy, surgery, or molecular targeted therapy within 4 weeks (or 5 drug half-lives, whichever is longer) prior to the first dose of the study drug; subjects with adverse events from previous treatments (excluding alopecia) that have not recovered to ≤CTCAE grade 1.
7. Subjects with clinically uncontrolled third-space effusion requiring puncture drainage or other local treatment prior to the first dose of the investigational drug.
8. Subjects with significant hemoptysis within 2 months before randomization, or hemoptysis of at least half a teaspoon (2.5 ml) per day.
9. Known hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism).
10. Subjects with active infection or unexplained fever >38.5°C during the screening period or prior to the first dose.
11. Subjects with a history of or current evidence of lung fibrosis, interstitial lung disease, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, or severely impaired lung function.
12. Subjects with congenital or acquired immune deficiencies (e.g., HIV infection) or active hepatitis (hepatitis B reference: HBV DNA exceeding the upper limit of normal; hepatitis C reference: HCV viral load or RNA exceeding the upper limit of normal).
13. Subjects who have used other investigational drugs or similar therapeutic agents within 4 weeks prior to the first dose or who have received radiotherapy or other local treatments within 2 weeks prior to the first dose and have not recovered from the adverse effects of such treatments.
14. Subjects with a history of or concurrent other malignancies (excluding cured basal cell carcinoma of the skin and cervical carcinoma in situ).
15. Subjects who may receive other systemic anti-tumor therapies during the study period.
16. Subjects who have received or are expected to receive live vaccines within 4 weeks prior to the first dose or during the study period.
17. Subjects with other factors that may lead to forced termination of the study as judged by the investigator, such as severe diseases (including mental disorders) requiring combined treatment, severe laboratory abnormalities, and family or social factors that may affect the safety of the subject or the collection of data and samples.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Progression-Free Survival (PFS) will be assessed from the date of enrollment until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 60 months
  Progression-Free Survival (PFS) will be assessed from the date of enrollment until the date of first documented disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate | ORR refers to the proportion of patients whose optimal response is complete or partial response, through study completion, an average of 2 years
  ORR refers to the proportion of patients whose optimal response is complete or partial response
Overall Survival | The time interval from enrollment to death from any cause, assessed up to 60 months
  The time interval from enrollment to death from any cause
Disease Control Rate | DCR refers to the proportion of patients whose optimal response is complete or partial response, or stable disease, through study completion, an average of 2 years
  DCR refers to the proportion of patients whose optimal response is complete or partial response, or stable disease
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Data will be recorded before each chemotherapy cycle, before and after radiotherapy, and every 3 months during the follow-up period, an average of 2 years
  Number of participants with adverse events and severe as assessed by CTCAE v5.0

OTHER OUTCOMES:
Biomarker | Biomarkers will be recorded before each chemotherapy cycle, before and after radiotherapy, and every 3 months during the follow-up period, an average of 2 years
  CD8A, PD-1, PD-L1, CD68, panCK, CD56, CD155, TIGIT, TMB, MSI, STING, et al

CONTACTS AND LOCATIONS:
Overall Officials: Peng Xie, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol